CLINICAL TRIAL: NCT05015335
Title: The Efficacy and Safety of Adalimumab for Inflammatory Flare Prevention in Non-infectious Anterior Pediatric Uveitis With Peripheral Vascular Leakage Compared With Methotrexate, a RCT Study
Brief Title: The Efficacy and Safety of Adalimumab in Non-infectious Anterior Pediatric Uveitis With Peripheral Vascular Leakage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25-ZS-3062
Record Dates: First submitted 2021-08-10; First posted 2021-08-20 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-07

CONDITIONS: Uveitis, Anterior; Adalimumab
Keywords: pheripheral retinal vasuclar leakage; adalimumab; methotrexate
MeSH Terms: conditions — Uveitis, Anterior | interventions — Adalimumab; Methotrexate

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center,open-lablel, interventional, randomizedcontrolled clinical trial that will be performed at the Ophthalmology Department, Peking Union Medical College Hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Adalimumab (Experimental): Adalimumab administered subcutaneously at 40mg every 2 weeks
  Interventions: Drug: Adalimumab
- Methotrexate (Active Comparator): Methotrexate given 10mg orally once a week.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Adalimumab — ADA 40mg q2w
  Other Names: ADA
  Arms: Adalimumab
Drug: Methotrexate — MTX 10mg qw
  Other Names: MTX
  Arms: Methotrexate

SUMMARY:
Children with anterior uveitis are prone to suffer from chronic recurrent course of intraocular inflammation and adverse effects of glucocorticosteroids (GCs) /immunomodulatory treatment (IMT) agents. The performance of adalimumab has been shown to be fairly favorable in treating refractory non-infectious uveitis. This study aims to assess the efficacy and safety of adalimumab for inflammatory flare prevention in non-infectious anterior pediatric uveitis with peripheral vascular leakage compared with methotrexate. Children weighed ≥ 30kg and aged between 4-16 years old with active chronic non-infectious anterior uveitis with peripheral retinal vascular leakage on ultra wildfield fluorescence fundus angiography (UWFFA) will be included. They will be treated with a predesigned inflammatory control regimen to reach inflammatory quiescence in 1 month. After that they will be treated with either MTX or adalimumab and regularly followed up for at least 6 months. The primary endpoint is treatment failure defined as any inflammatory fare with anterior chamber cell count grading increased from 0 to 1. Secondary endpoints are best corrected visual acuity (BCVA), inflammation parameters (keratic precipitates, vitreous haze grades), extent of vascular leakage, frequency of topical steroid eyedrops, systemic immunosuppressive drug load, and adverse events.

DETAILED DESCRIPTION:
This is a prospective, single-center, interventional, randomized, non-blinded, controlled clinical trial that will be performed at the Ophthalmology Department, Peking Union Medical College Hospital.

Children with active noninfectious anterior uveitis demonstrating peripheral vascular leakage on UWFFA and meet the selection criteria will be randomly assigned to treatment group or control group.

Both groups will be treated with a predesigned plan for the active inflammation. At one month or when patients' ocular inflammation gets controlled to 0.5+ cell in the anterior chamber, whichever comes later, patients in the treatment group will be given adalimumab subcutaneously at 40mg every 2 weeks, patients in the control group will be given methotrexate10mg orally once a week.

Follow-up visits will be scheduled every two weeks at the run-in period and the first month after randomization, and every month from the second to the sixth month.

The primary endpoint is treatment failure defined as any inflammatory fare with anterior chamber cell count grading increased from 0 to 1.

Secondary endpoints are best corrected visual acuity (BCVA), inflammation parameters (keratic precipitates, vitreous haze grades), extent of vascular leakage, frequency of topical steroid eyedrops, systemic immunosuppressive drug load, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Children with noninfectious uveitis aged between 4-16, weight ≥ 30kg.
2. Uveitis resistant to well conducted topical steroid therapy for three months, or uveitis resistant to well conducted 0.1% prednisolone twice a day for one month
3. Retina peripheral vascular leakage demonstrated by UWFFA at the time of inclusion.

Exclusion Criteria:

1. Any contraindication to administration of immunosuppressive therapy (active tuberculosis, immune deficit, opportunistic infection, other severe chronic disease).
2. Previous diagnosis or signs of demyelinating disease of the central nervous system.
3. Children unable to cooperate with examinations and follow-up.
4. Positive allergy skin test when conducting fluorescence fundus angiography.
5. Diffuse vascular leakage, macula edema or any retina lesions demonstrated by UWFFA.
6. History of oral immunosuppressive drug treatment within 2 months
7. History of biological treatment within 2 months
8. History of triamcinolone acetonide subconjunctival/intraocular injection within 3 months
9. Current topical steroid use more than six times per day
10. History of eye surgery within 3 months.
11. Eye complications that interfere with fundus observation.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Uveitis flare | At 6 months' follow-up visit
  Uveitis flare is defined as anterior chamber cell count grading increased from 0 to 1.
  The grading method is in accordance with SUN criteria. Anterior chamber cell count was scored according to Standardization of Uveitis Nomenclature (SUN) criteria

SECONDARY OUTCOMES:
Extent of peripheral vascular leakage | At 6 months' follow-up visit
  Vascular leakage was quantified based on the method developed by the Angiography Scoring for Uveitis Working Group (ASUWOG), in which vascular leakage in the posterior pole and in each peripheral quadrant was scored 1 if limited and scored 2 if diffuse. Total maximum score will 8 since leakage in the posterior pole will be excluded in this study.
Keratic precipitates | At 6 months' follow-up visit
  Keratic precipitates was recorded in a dichotomous method.
Vitreous haze | At 6 months' follow-up visit
  Vitreous haze will graded as the same method of anterior chamber cell, the slit lamp will be pushed forward to the vitreous to observe vitreous haze.
Best corrected visual acuity (BCVA) | At 6 months' follow-up visit
  BCVA was transformed into logMar form
Adverse events | through study completion, an average of 6 months
  Adverse events included the infectious events and laboratory parameter abnormalities.
frequency of topical steroid eyedrops if any inflammatory flare happens. | At 6 months' follow-up visit
  Different GCs eye drops are transformed into equivalent 1% prednisolone for analysis.
Systemic immunomodulatory therapy (sIMT, including GCs and immunosuppressive drugs)load at the 6-month follow-up visit if any inflammatory flare ever happens. | At 6 months' follow-up visit
  sIMT load is transformed into a quantizable score based on prior studies in uveitis.

CONTACTS AND LOCATIONS:
Overall Officials: Meifen Zhang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking University Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
If other researcher needs the IPD. Please contact songhang_pumch@163.com

REFERENCES:
- [Background] Agrawal R, Agarwal A, Jabs DA, Kee A, Testi I, Mahajan S, McCluskey PJ, Gupta A, Palestine A, Denniston A, Banker A, Invernizzi A, Fonollosa A, Sharma A, Kumar A, Curi A, Okada A, Schlaen A, Heiligenhaus A, Kumar A, Gurbaxani A, Bodaghi B, Islam Shah B, Lowder C, Tappeiner C, Muccioli C, Vasconcelos-Santos DV, Goldstein D, Behra D, Das D, Makhoul D, Baglivo E, Denisova E, Miserocchi E, Carreno E, Asyari F, Pichi F, Sen HN, Uy H, Nascimento H, Tugal-Tutkun I, Arevalo JF, Davis J, Thorne J, Hisae Yamamoto J, Smith J, Garweg JG, Biswas J, Babu K, Aggarwal K, Cimino L, Kuffova L, Agarwal M, Zierhut M, Agarwal M, De Smet M, Tognon MS, Errera MH, Munk M, Westcott M, Soheilian M, Accorinti M, Khairallah M, Nguyen M, Kon OM, Mahendradas P, Yang P, Neri P, Ozdal P, Amer R, Lee R, Distia Nora R, Chhabra R, Belfort R, Mehta S, Shoughy S, Luthra S, Mohamed SO, Chee SP, Basu S, Teoh S, Ganesh S, Barisani-Asenbauer T, Guex-Crosier Y, Ozyazgan Y, Akova Y, Habot-Wilner Z, Kempen J, Nguyen QD, Pavesio C, Gupta V; Collaborative Ocular Tuberculosis Study (COTS) Group. Standardization of Nomenclature for Ocular Tuberculosis - Results of Collaborative Ocular Tuberculosis Study (COTS) Workshop. Ocul Immunol Inflamm. 2020 Sep 30;28(sup1):74-84. doi: 10.1080/09273948.2019.1653933. Epub 2019 Dec 10. PMID 31821096
- [Background] Nussenblatt RB, Peterson JS, Foster CS, Rao NA, See RF, Letko E, Buggage RR. Initial evaluation of subcutaneous daclizumab treatments for noninfectious uveitis: a multicenter noncomparative interventional case series. Ophthalmology. 2005 May;112(5):764-70. doi: 10.1016/j.ophtha.2004.12.034. PMID 15878055
- [Background] Tugal-Tutkun I, Herbort CP, Khairallah M; Angiography Scoring for Uveitis Working Group (ASUWOG). Scoring of dual fluorescein and ICG inflammatory angiographic signs for the grading of posterior segment inflammation (dual fluorescein and ICG angiographic scoring system for uveitis). Int Ophthalmol. 2010 Oct;30(5):539-52. doi: 10.1007/s10792-008-9263-x. Epub 2008 Sep 16. PMID 18795232
- [Result] Ramanan AV, Dick AD, Jones AP, McKay A, Williamson PR, Compeyrot-Lacassagne S, Hardwick B, Hickey H, Hughes D, Woo P, Benton D, Edelsten C, Beresford MW; SYCAMORE Study Group. Adalimumab plus Methotrexate for Uveitis in Juvenile Idiopathic Arthritis. N Engl J Med. 2017 Apr 27;376(17):1637-1646. doi: 10.1056/NEJMoa1614160. PMID 28445659
- [Derived] Song H, Zhao C, Zhang Y, Li D, Qian Y, Gao F, Xiao J, Zhang M. Efficacy and safety of adalimumab for inflammatory flare prevention in paediatric non-infectious anterior uveitis with peripheral retinal vascular leakage: a study protocol for a single-centre, randomised controlled trial. BMJ Open. 2022 Dec 7;12(12):e062211. doi: 10.1136/bmjopen-2022-062211. PMID 36600374